CLINICAL TRIAL: NCT06246877
Title: Effect of Virtual Reality on Pain and Fear Level During Kirschner Wires (K-Wires) Removal and Dressing in Children
Brief Title: Virtual Reality on Pain and Fear Level During Kirschner Wires (K-Wires) Removal in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Esra TURAL BUYUK, Assoc Prof, Ondokuz Mayıs University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: K Teli
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Fear of Pain
Keywords: child; Kirschner Wires; pain; fear; Virtual reality
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- virtual reality applied group (Experimental): Before the K-wire is removed and dressed, the three-dimensional video that the child likes and wants to watch will be placed on virtual reality glasses and attached to the child.
  During the procedure, the child will be allowed to watch videos through virtual reality glasses.
  Interventions: Behavioral: virtual reality applied group
- control group (No Intervention): During the removal and dressing of the wire, the child's attention will be diverted by asking some questions (where she lives, the name of the school she attends, what grade she attends, etc.).

INTERVENTIONS:
Behavioral: virtual reality applied group — Before the K-wire is removed and dressed, the three-dimensional video that the child likes and wants to watch will be placed on virtual reality glasses and attached to the child.
  During the procedure, the child will be allowed to watch videos through virtual reality glasses.
  Arms: virtual reality applied group

SUMMARY:
This study will be conducted to examine the effect of virtual reality applied during K-wire removal and dressing on the pain and fear levels that develop due to the procedure in children aged 7-12 years who apply to the orthopedic outpatient clinic.

DETAILED DESCRIPTION:
Technology-based methods have now begun to be used to control anxiety and prevent pain that may occur before, during and after diagnosis and treatment procedures in children.

Virtual reality (VR), which is among the technological products, can be used in non-pharmacological methods as well as pharmacological methods.

It has been observed that VR, especially in children, creates an analgesic effect by mainly distracting the pain centers in the brain and evokes positive emotions with an anxiolytic effect.Since children do not want to see the procedures to be performed on them, virtual reality used during the procedure is one of the methods of diverting attention from the environment they are in. This study will be conducted to examine the effect of virtual reality applied during K-wire removal and dressing on the pain and fear levels that develop due to the procedure in children aged 7-12 years who apply to the orthopedic outpatient clinic.

ELIGIBILITY:
Inclusion Criteria:

* Being a child between the ages of 7-12 who will have the K wire removed
* The child is not using glasses
* The child must be at a cognitive development level that can respond to video selection.

Exclusion Criteria:

* Having a disease that causes chronic pain
* The child must have used medication that would have an analgesic effect in the last 24 hours before the application.
* The child is wearing glasses
* The child has a mental or neurological disability

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Wong-Baker Faces Pain Scale | The "Wong-Baker Faces Pain Scale" will be scored 5 minutes before K-wire removal and dressing. It will be evaluated again by scoring the "Wong-Baker Faces Pain Scale" 5 minutes after the K-wire removal and dressing.
  It is suitable for ages three and above. The pain level of the faces on the scale is explained to the child: "Face 0" indicates that there is no pain and is very happy. "Face 2" has some pain. "Face 4" has slightly more pain. "Face 6" has more pain. The pain of "Face 8" is quite severe. The pain of "Face 10" is unbearable.

SECONDARY OUTCOMES:
Children's Fear Scale | "Child Fear Scale" scoring will be done 5 minutes before K-wire removal and dressing. It will be evaluated again by scoring the "Child Fear Scale" 5 minutes after the K-wire removal and dressing.
  The scale is a scale that evaluates between 0 and 4, consisting of showing five drawn facial expressions ranging from neutral expression (0 = no anxiety) to scared face (4 = severe anxiety).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Ondokuz Mayıs University Faculty of Health Sciences, Samsun, Atakum
  - Bafra State Hospital, Samsun